CLINICAL TRIAL: NCT02658019
Title: Phase II Study of Pembrolizumab (Keytruda®) in Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Pembrolizumab (Keytruda) in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynn Feun, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Lynn Feun, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20151049
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Advanced Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab in Advanced HCC (Experimental): Patients will be treated in three-week cycles, with intravenous (IV) administration of 200 mg of pembrolizumab on day 1 of each 3-week cycle. Trial therapy will last until withdrawal of consent, disease progression and/or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patients will be treated in three-week cycles, with intravenous (IV) administration of 200 mg of pembrolizumab on day 1 of each 3-week cycle.
  Other Names: Keytruda; MK-3475

SUMMARY:
This is a single-arm phase II trial of Pembrolizumab (Keytruda) in patients with advanced, unresectable hepatocellular carcinoma. The primary objective is to assess its therapeutic efficacy in patients with unresectable hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have diagnosis of advanced hepatocellular cancer (HCC) by one of the following:

   * Histopathology
   * Elevated serum alpha-fetoprotein (AFP) >400 ng/ml and findings on magnetic resonance imaging (MRI) or computed tomography (CT) scans characteristic of HCC
   * Findings on triple phase MRI or CT scans characteristic of HCC in patients with cirrhosis and tumors at least 1 cm or greater, without a curative treatment option (transplant, resection, or ablation).
2. Measurable disease as defined by RECIST v1.1 (provided in Section 14.0).
3. Radiographic progression on previously treated areas (as defined by RECIST v1.1).
4. Subject refusal for sorafenib treatment or intolerance to sorafenib are also allowed (intolerance is defined as ≥ 28 days of sorafenib (not necessarily consecutive) or ≥grade 3 toxicity due to sorafenib which does not resolve with appropriate supportive care).
5. Patients should have failed at least one prior systemic therapy regimen which could include sorafenib. Patients may have progressed on sorafenib, been intolerant of, or refused sorafenib. Patients who are documented to refuse systemic chemotherapy or sorafenib are also eligible. No limit to prior systemic therapy. Prior locoregional therapy such as surgery, radiofrequency ablation or transarterial chemoembolization are also allowed, provided that progression has been documented after these therapies, and ≥4 weeks have elapsed since the last therapy; (these will not be counted as systemic therapy).
6. Child-Pugh Classification with score ≤ 7 points. See Appendix G for criteria.
7. Age ≥ 18 years
8. Estimated life expectancy, in the judgement of the Investigator, of at least ≥ 12 weeks.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. See Appendix C.
10. Adequate bone marrow function as defined below:

    * absolute neutrophil count (ANC) ≥ 1.2 x 10^9/L,
    * platelets (PLT) ≥ 50 x 10^9/L
11. Adequate liver function as defined below:

    * serum bilirubin < 2 mg/dl
    * Aspartate transaminase (AST/SGOT) ≤ 5 x upper limit of normal (ULN),
    * Alanine transaminase (ALT/SGPT) ≤ 5 x ULN
12. Adequate coagulation as defined by:

    * serum prothrombin time (PT) ≤ 16 seconds
13. Adequate renal function as defined by one of the following:

    * serum Creatinine ≤ 1.5 x ULN OR
    * (measured or calculated) Creatinine clearance ≥ 60 mL/min for patients with serum creatinine levels > 1.5 x ULN.
14. Suitable venous access to allow for all study-related blood sampling.
15. Female subject of childbearing potential (CBP) must have a negative urine or serum pregnancy within 3 days prior to receiving the first dose of study medication.
16. Females of child bearing potential that are sexually active must agree to either practice 2 medically accepted highly effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 120 days after the last dose of study drug. See Appendix H for protocol-approved highly effective methods of contraceptive combinations. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
17. Negative test for pregnancy is required of females of child-bearing potential; A female of child bearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

    * has not undergone a hysterectomy or bilateral oophorectomy; or
    * has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months or 730 days).
18. Conception while on treatment must be avoided
19. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
20. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
2. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 years prior to the first dose of trial treatment.
3. Major surgical procedure within 28 days prior to enrollment. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
4. Any unresolved toxicity > CTCAE grade 2 despite optimal care/support, from previous anti-cancer therapy, within 28 days prior to first dose of study drug. [Exceptions: Alopecia and ≤grade 2 neuropathy.]
5. Prior therapy with an anti-Programmed Death (PD)-1, anti-PD-Ligand-(L)-1, or anti-PD-L2 agent.
6. Receipt of anti-cancer monoclonal antibody within 4 weeks prior to first dose of study drug.
7. Prior treatment with any other chemotherapy, radiotherapy, immunotherapy, or anticancer drug, agent or biologic within 4 weeks prior to first dose of study drug.
8. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
9. Receipt of any other investigational agents for their cancer ≤4 weeks of the first dose of study treatment.
10. Known history of active Bacillus Tuberculosis (TB).
11. Known history of, or any evidence of active, non-infectious pneumonitis or has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Known history of Human Immunodeficiency Virus (HIV), HIV-1/2 antibodies.
13. Known hypersensitivity to pembrolizumab or any of its excipients.
14. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. [Exception: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging, for at least 4 weeks prior to the first dose of study drug and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not apply to carcinomatous meningitis which is excluded regardless of clinical stability.]
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 120 days after the last dose of trial treatment.
16. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
17. Has a known additional malignancy that is progressing or requires active treatment. [Exception: Basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.]
18. Any other serious medical or psychiatric illness/condition likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
19. Treatment for active hepatitis C virus (HCV) within 60 days of study entry. [Note: Untreated HCV positive subjects are eligible, and if stable on pembrolizumab for 6 months after study entry, consideration may be given to starting anti-HCV therapy, at the discretion of the treating Investigator.]
20. HCC patients with evidence of prior hepatitis B virus (HBV) must fulfill the following criteria in order to be eligible for the study: HBV viral load (VL) <100 IU/mL before study enrollment, and subjects with active HBV need to be on anti-HBV suppression ≥3 months, throughout treatment and for 6 months after.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Feun, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feun LG, Li YY, Wu C, Wangpaichitr M, Jones PD, Richman SP, Madrazo B, Kwon D, Garcia-Buitrago M, Martin P, Hosein PJ, Savaraj N. Phase 2 study of pembrolizumab and circulating biomarkers to predict anticancer response in advanced, unresectable hepatocellular carcinoma. Cancer. 2019 Oct 15;125(20):3603-3614. doi: 10.1002/cncr.32339. Epub 2019 Jun 28. PMID 31251403
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab in Advanced HCC
Started | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) in Study Participants
Description: Disease control rate (DCR) will be calculated per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, as the percentage of patients with best overall response to protocol therapy of either complete response (CR), partial response (PR) or stable disease (SD) that is maintained for at least 8 weeks.
  Per Response Evaluation Criteria in Sold Tumors Criteria (RECISTv1.1)for target lesions and assessed by MRI or CT: Complete response(CR),Disappearance of all target lesions; Partial response(PR),>=30% decrease in sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 28
percentage of participants | 46 [27.5 to 66.1]

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: The safety of Pembrolizumab in HCC patients as measured by the incidence of treatment-related adverse events, including serious adverse events (SAEs), in study participants using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, per physician discretion. The number of participants experiencing toxicity attributed by treating physician as definitely, probably and possibly-related to study treatment will be reported.
Time Frame: Up to 2 years
Population: One participant experienced two SAEs; one with attribution of possible relation, and the second with probable relation to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 29
Participants
  SAEs with Attribution of Definite Relation | 0
  SAEs with Attribution of Possible relation | 6
  SAEs with Attribution of Probable Relation | 2
  AEs with Attribution of Definite Relation | 0
  AEs with Attribution of Possible Relation | 26
  AEs with Attribution of Probable Relation | 16

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment .
Time Frame: Up to 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 28
months | 4.5 [2 to 7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive).
Time Frame: Up to 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 28
months | 11 [7 to 19]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) will be defined as the percentage of the patients with a confirmed complete or partial response (CR or PR),by MRI or CT scan as per RECIST 1.1 criteria. Complete response (CR), Disappearance of all target lesions; Partial response (PR), >=30% decrease in sum of the longest diameter of target lesions; Overall response (OR) = (CR+PR.)Scans and assessments are performed every 9 weeks while on treatment up to 2 years if stable/responding, or up until time of disease progression.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 28
percentage of participants | 32 [15.9 to 52.4]

6. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) will be defined as the elapsed time from documented tumor response to documented disease progression.
Time Frame: Up to 3 Years
Population: Median duration of response was not achieved for the participants by the end of study participation at the 3-year follow up visit.
Arm/Group | Pembrolizumab in Advanced HCC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 25 months
Description: Only treatment-emergent adverse events and serious adverse events are reported for this protocol. A treatment-emergent adverse event and serious adverse events (TEAE) are defined as any event that begins or worsens after the start of protocol treatment with a treating physician attribution of definite, probable or possible relation to treatment. One participant experienced two SAEs; one with attribution of possible relation, and the second with probable relation to study treatment.
Arm/Group | Pembrolizumab in Advanced HCC
All-Cause Mortality (participants affected / at risk) | 9/29
Serious Adverse Events (participants affected / at risk) | 7/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab in Advanced HCC (N=29)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab in Advanced HCC (N=29)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (16)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (12)
Blood bilirubin increased (Investigations) | 9 (20)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (26)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Peri-orbital tenderness (Eye disorders) | 1 (1)
Fatigue (General disorders) | 11 (15)
Fever (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 6 (15)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Localized edema (General disorders) | 1 (1) — Bilateral Lower Limb Edema
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow tenderness (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Neutrophil count decreased (Investigations) | 4 (9)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Papulopustular rash (Infections and infestations) | 2 (3)
Platelet count decreased (Investigations) | 5 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Nail Change (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3)
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02658019/Prot_SAP_000.pdf